CLINICAL TRIAL: NCT01638988
Title: Clomifene Citrate Versus Metformin in First-line Treatment of Infertility in Patients With Polycystic Ovary Syndrome (PCOS) and a Resistance to Insulin. Randomised Controlled Study
Brief Title: Clomifene Citrate Versus Metformin in First-line Treatment of Infertility in Patients With Polycystic Ovary Syndrome and a Resistance to Insulin
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Previous studies have been done regarding same condition
Sponsor: Clinique Ovo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OVO-12-17
Record Dates: First submitted 2012-07-09; First posted 2012-07-12 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Polycystic Ovary Syndrome; Insulin Resistance
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance | interventions — Metformin; Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Experimental)
  Interventions: Drug: Metformin
- Clomiphene Citrate (Active Comparator)
  Interventions: Drug: Clomiphene citrate

INTERVENTIONS:
Drug: Metformin — 1. cycle 2000 mg of Metformin : Day 1 to day 30; beginning with 1/2 tablet by day with an increasing until 4 pills by day
  2. to 6 cycle 2000 mg of Metformin : Day 1 ot day 30; 4 pills of Metformin by day Positive pregnancy test : 4 pills of Metformin by day until 12 weeks of pregnancy
  Arms: Metformin
Drug: Clomiphene citrate — Cycle 1: Day 3 to day 7; 50 mg; 1 tablet of Clomiphene Citrate by day Cycle 2: Day 3 to day 7; 100 mg; 1 tablet of Clomiphene Citrate two times a day Cycle 3 to 6 : Day 3 to day 7; 150 mg; 1 tablet of Clomiphene Citrate 3 times a day
  Arms: Clomiphene Citrate

SUMMARY:
The results of studies conducted until now does not determine what the best way to treat infertility in the first line with patients with Polycystic ovary syndrome (PCOS). This study objective is to determine the best treatment for such patients. The long-term consequence health of women with PCOS are multiple. The woman with PCOS has a risk of developing metabolic diseases, heart diseases, diabetes Type II or anovulatory infertility. The insulin resistance plays an important role in all this medical condition. Clomiphene Citrate (CC) remains the first line treatment to induce ovulation in women with PCOS and anovulatory infertility.

ELIGIBILITY:
Inclusion Criteria:

* Women aged from 18 to 35
* Infertility for a period of a year or more or 6 month of irregular menstrual cycle
* PCOS under the Rotterdam criteria
* Insulin resistance HOMA-IR > 2.5
* Normal semen analysis values
* Normal values of the following blood analysis: FSH, LH, Estradiol, AMH, TSH, Prolactine, Fasting glucose level, hemoglobin A1C, AST, ALT, alkaline phosphatase, SHBG, 17OH progesterone, DHEAS, Androstenedione, total testosterone, LDL, HDL, total cholesterol, Triglycerides, oral glucose tolerance test

Exclusion Criteria:

* Tubular factor
* Normal ovarian reserve
* Prior use of CC or Metformin, hypoglycemic agents, glucocorticoids, anti-androgen, weight-loss agent or oral contraceptives in the past 6 months
* Neoplasia
* BMI > 35
* Renal, hepatic or cardiac failure
* Lactic, acidosis antecedent

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Biochemical pregnancy | 1 month
  Rate of biochemical pregnancy

SECONDARY OUTCOMES:
Ovulation rate | 1 month
  Ovulation rate
Live birth rate | 6 months
Spontaneous abortion rate | 6 months
BMI and waist size changing | 6 months
Insulin resistance changing | 6 months
AMH correlation/variation in function of Metformin | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Kadoch, Dr, Principal Investigator — Clinique Ovo
Locations (1):
- Clinique Ovo, Montreal, Quebec, Canada